CLINICAL TRIAL: NCT04356027
Title: Validation of OCT-based FUnctional diagnoSIs of corONary Stenosis (FUSION)
Brief Title: FUnctional diagnoSIs of corONary Stenosis (FUSION)
Acronym: FUSION
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10331
Record Dates: First submitted 2020-04-20; First posted 2020-04-21 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: Virtual Flow Reserve (VFR); Optical Coherence Tomography (OCT); Fractional Flow Reserve (FFR); Percutaneous Coronary Intervention (PCI); OPTIS System; Dragonfly; PressureWire X
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care: Angiography, OCT, FFR, and VFR: Patients will have Pre-OCT Angiography, OCT pullbacks, a FFR measurement and a VFR analysis
  Interventions: Procedure: ICA (Invasive Coronary Angiography); Procedure: OCT; Procedure: FFR; Other: VFR Analysis

INTERVENTIONS:
Procedure: ICA (Invasive Coronary Angiography) — Patients will undergo a Pre-PCI Angiography
Procedure: OCT — OCT pullback images will be collected pre-PCI and (optional) post-PCI procedure
Procedure: FFR — FFR will be measured
Other: VFR Analysis — VFR will be calculated offline using the OCT pullback images

SUMMARY:
The purpose of the FUSION study is to validate the diagnostic performance of Virtual Flow Reserve (VFR) by comparing it against a reference standard, fractional flow reserve (FFR).

DETAILED DESCRIPTION:
This study is a single-arm, prospective, multi-center study collecting OCT pullback images of lesions pre-percutaneous coronary intervention (PCI) and (optional) post-PCI procedure, and the corresponding pressure tracings and physiology indices. Up to 30 centers in the US will enroll approximately 310 patients. The expected duration of enrollment is approximately 15 months. The total duration of the clinical investigation is expected to be approximately 27 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient provides written informed consent
* Scheduled for clinically indicated coronary catheterization with the intent to perform physiologic assessment to guide physician clinical course (in lesions with visual % diameter stenosis 40-90%), if clinically indicated
* Subject is undergoing invasive FFR with Adenosine (high-dose intra-coronary (IC) [200 μg for the left and or 100 μg for the right coronary artery] or 140 μg/kg/min for intravenous (IV)) used as hyperemic stimulus
* Clinical presentation with or history of stable angina, unstable angina, or silent ischemia (defined as abnormal stress test or abnormal invasive physiology assessment) that has led to the procedure

General Exclusion Criteria:

* Prior history of myocardial infarction (MI) in the target vessel
* Presence of acute ST Elevation Myocardial Infarction (STEMI)
* Culprit vessel of Non-ST Elevation Myocardial Infarction (NSTEMI)
* TIMI flow < Grade 3 at baseline or visible thrombus
* Prior history of coronary artery bypass grafting (CABG)
* Prior heart transplant
* Severe valvular heart disease or history of valve repair or replacement
* Prior history of PCI with stent in target vessel, or target vessel involves in-stent restenosis.
* Target coronary vessel is supplied by major collaterals or is supplying major collaterals to a CTO (chronic total occlusion)
* CTO in the target vessel
* Severe diffuse disease observed in target vessel defined as the presence of diffuse, serial gross luminal irregularities present in the majority of the coronary tree
* Presence of myocardial bridge (MB), regardless of vessel location
* Contraindication for FFR examination or administration of vasodilators
* Known LVEF ≤45%
* Target lesion involves Left Main coronary artery or ostial right coronary artery
* Known renal insufficiency (eGFR < 30 ml/kg/m^2 or serum creatinine ≥ 2.5 mg/dL) unless patient is on dialysis
* Heart Failure NYHA Class III or IV
* Subject is pregnant (For a female subject of childbearing potential, a pregnancy test must be performed within 14 days (≤14 days) prior to the index procedure per site standard test)
* Subject has or had active COVID-19 symptoms and/or a positive test result within the prior 2 months
* Participation in another clinical study of an investigational drug or device
* Presence of aneurysm in the target vessel

Imaging and Pressure Tracing Exclusion Criteria:

* Artifact in pre-PCI OCT for the target lesion or in the event of multiple target lesions, artifact in pre-PCI OCT for ALL target lesions
* Target lesion requires any preparation (including but not limited to balloon dilatation, atherectomy, etc.) prior to pre-PCI OCT and physiology measurement, or in case of multiple target lesions, ALL target lesions require-any preparation (including but not limited to balloon dilatation, atherectomy, etc.) prior to pre-PCI OCT and physiology measurement
* Severe vessel tortuosity or calcification in the target vessel such that it is unlikely that the OCT catheter can be delivered
* Target lesion not imaged by OCT or in the event of multiple target lesions, ALL target lesions not imaged by OCT
* Pressure drift of > 0.03; i.e. Pd and Pa ratio value < 0.97 or > 1.03, unless physiology measurements are repeated after re-equalization
* Target lesion or significant CAD beyond 60mm from coronary ostium; i.e. not able to clearly image and capture all disease segment with OCT in 1 run
* Incorrectly done or unsuccessful catheter purge and/or contrast flush
* Presence of plaque rupture and/or intravascular hematoma in target vessel (visual % diameter stenosis ≥ 40%)
* Inability to receive intracoronary nitroglycerin prior to OCT or FFR
* Use of flush media other than radiographic contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll male and female subjects from the general interventional cardiology population.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Jeremias, MD, Principal Investigator — St. Francis Hospital,Roslyn,NY, United States
Locations (28):
- United States (28):
  - Heart Center Research, LLC., Huntsville, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - VA Palo Alto Medical Center, Palo Alto, California
  - UCLA Medical Center Santa Monica, Santa Monica, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - The Cardiac & Vascular Institute Research Foundation, LLC, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mercy Hospital, Coon Rapids, Minnesota
  - St. Patrick Hospital, Missoula, Montana
  - New York University Hospital, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - VA Medical Center Durham, Durham, North Carolina
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Austin Heart, Austin, Texas
  - University of Texas Medical Branch (UTMB), Galveston, Texas
  - Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeremias A, Maehara A, Matsumura M, Shlofmitz RA, Maksoud A, Akasaka T, Bezerra HG, Fearon WF, Samady H, Samuels B, Rapkin J, Gopinath A, Teraphongphom NT, Buccola J, Ali ZA. Optical Coherence Tomography-Based Functional Stenosis Assessment: FUSION-A Prospective Multicenter Trial. Circ Cardiovasc Interv. 2024 Apr;17(4):e013702. doi: 10.1161/CIRCINTERVENTIONS.123.013702. Epub 2024 Mar 25. PMID 38525609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 312 subjects with a total of 315 vessels from 27 sites. After being reviewed for quality by the core laboratory, 224 pre-PCI and 42 post-PCI vessels from 224 subjects remained for the endpoints analysis.
Units Other Than Participants: vessels
Groups:
- Standard of Care: Angiography, OCT, FFR, and VFR: This is a single arm study. Patients will have Pre-OCT Angiography, OCT pullbacks, a FFR measurement and a VFR analysis
  ICA (Invasive Coronary Angiography): Patients will undergo a Pre-PCI Angiography
  OCT: OCT pullback images will be collected pre-PCI and (optional) post-PCI procedure
  FFR: FFR will be measured
  VFR Analysis: VFR will be calculated offline using the OCT pullback images
Period: Overall Study
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Started | 224; 266 vessels
Pre PCI | 224; 224 vessels
Post PCI | 224; 42 vessels
Completed | 224; 266 vessels
Not Completed | 0; 0 vessels

BASELINE CHARACTERISTICS:
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Number analyzed (Participants) | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 191
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 224
Hyperlipidemia [Number; unit: participants] | 186
Hypertension [Number; unit: participants] | 182

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Virtual Flow Reserve (VFR) Against Fractional Flow Reserve (FFR)
Description: Sensitivity and specificity of the VFR compared with FFR each of which will be tested against a prespecified performance goal. FFR with a binary cut-off of 0.80 will be used as the reference standard for comparison.
  FFR or VFR value ≤ 0.80 will be considered positive (ischemia-causing), and FFR or VFR value > 0.80 will be considered negative (non-ischemia-causing).
  Sensitivity is defined as the percentage of VFR positive lesions, in the group of FFR positive lesions.
  Sensitivity=TP/(TP+FN) x 100%, where TP denotes the number of True Positives (both VFR and FFR positive) and FN denotes the number of False Negatives (VFR negative but FFR positive).
  Specificity is defined as the percentage of VFR negative lesions in the group of FFR negative lesions.
  Specificity=TN/(TN+FP) x 100%, where TN denotes the number of True Negatives (both VFR and FFR negatives) and FP denotes the number of False Positives (VFR positive but FFR negative).
Time Frame: Baseline (pre-procedure) and immediately post-procedure
Population: The primary analysis population included vessels in enrolled subjects having acceptable OCT pullbacks and pressure tracings for computing both the VFR and FFR indices. This is a single-arm study, so there is no data to report per arm, only data collected at different time points throughout the study.
Measure: Number; unit: vessels
Units Other Than Participants: Vessels
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Number analyzed (Participants) | 224
Number analyzed (Vessels) | 266
vessels
  Sensitivity: number analyzed (Vessels) | 102
  Sensitivity | 82
  Specificity: number analyzed (Vessels) | 164
  Specificity | 136

2. Secondary Outcome: Overall Diagnostic Accuracy
Description: Overall diagnostic accuracy is defined as the proportion of correctly classified lesions among all lesions.
  Overall Diagnostic Accuracy= (TP+TN)/(TP+TN+FP+FN) x 100%, where TP denotes the number of True Positives, FN denotes the number of False Negatives, TN denotes the number of True Negatives, and FN denotes the number of False Negatives.
Time Frame: Baseline (pre-procedure) and immediately post-procedure
Population: as for outcome 1
Measure: Number; unit: vessels
Units Other Than Participants: Vessels
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Number analyzed (Participants) | 224
Number analyzed (Vessels) | 266
vessels | 218

3. Secondary Outcome: Positive Predictive Value (PPV) and Negative Predictive Value (NPV)
Description: PPV is defined as the proportion of lesions with the disease and with a positive test result among the group of lesions with a positive test result.
  PPV= TP/(TP+FP) x 100%, where TP denotes the number of True Positives and FP denotes the number of False Positives.
  NPV is defined as the proportion of lesions without the disease and with a negative test result among the group of lesions with negative test results.
  NPV= TN/(TN+FN) x 100%, where TN denotes the number of True Negatives and FN denotes the number of False Negatives.
Time Frame: Baseline (pre-procedure) and immediately post-procedure
Population: as for outcome 1
Measure: Number; unit: vessels
Units Other Than Participants: Vessels
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Number analyzed (Participants) | 224
Number analyzed (Vessels) | 266
vessels
  PPV number analyzed: number analyzed (Vessels) | 110
  PPV number analyzed | 82
  NPV number analyzed: number analyzed (Vessels) | 156
  NPV number analyzed | 136

4. Secondary Outcome: Correlation Between VFR and FFR
Description: The correlation between VFR and FFR will be estimated as the R^2 correlation coefficient from the simple linear regression model using VFR value as the independent variable and FFR as the dependent variable.
Time Frame: Baseline (pre-procedure) and immediately post-procedure (post-procedure)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Vessels
Groups:
- Standard of Care: Angiography, OCT, FFR, and VFR: This is a single arm study. Patients will have Pre-OCT Angiography, OCT pullbacks, a FFR measurement and a VFR analysis.
  ICA (Invasive Coronary Angiography): Patients will undergo a Pre-PCI Angiography.
  OCT: OCT pullback images will be collected pre-PCI and (optional) post-PCI procedure.
  FFR: FFR will be measured.
  VFR Analysis: VFR will be calculated offline using the OCT pullback images.
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Number analyzed (Participants) | 224
Number analyzed (Vessels) | 266
correlation coefficient | 0.4992 [0.4105 to 0.5807]

5. Secondary Outcome: Area Under Curve (AUC) Against FFR
Description: AUC will be estimated as the area under the ROC curve. ROC curve will be constructed using specificity on the x-axis and sensitivity on the y-axis. Sensitivity and specificity are calculated at various values of VFR and FFR, and the AUC curve will be drawn using logistic regression.
Time Frame: Baseline (pre-procedure) and immediately post-procedure (post-procedure)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Vessels
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
Number analyzed (Participants) | 224
Number analyzed (Vessels) | 266
probability | 0.8790 [0.8380 to 0.9199]

ADVERSE EVENTS:
Time Frame: Immediately post-procedure
Description: The study enrolled a total of 312 subjects with a total of 315 vessels from 27 sites. After being reviewed for quality by the core laboratory, only 224 pre-PCI and 42 post-PCI vessels from 224 subjects remained for the endpoints analysis
Arm/Group | Standard of Care: Angiography, OCT, FFR, and VFR
All-Cause Mortality (participants affected / at risk) | 0/312
Serious Adverse Events (participants affected / at risk) | 5/312
Other Adverse Events (participants affected / at risk) | 3/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care: Angiography, OCT, FFR, and VFR (N=312)
Vascular Dissection (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Vessel Perforation (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care: Angiography, OCT, FFR, and VFR (N=312)
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Vascular Dissection (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT04356027/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04356027/SAP_001.pdf